CLINICAL TRIAL: NCT02471196
Title: Efficacy of ORM-12741 on Agitation/Aggression Symptoms in Patients With Alzheimer's Disease: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Multicentre Study of 12 Weeks
Brief Title: Efficacy of ORM-12741 on Agitation/Aggression Symptoms in Alzheimer's Disease
Acronym: Nebula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3098012
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ORM-12741

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ORM-12741 low dose (Experimental): ORM-12741 low dose twice a day for 12 weeks.
  Interventions: Drug: ORM-12741
- ORM-12741 high dose (Experimental): ORM-12741 high dose twice a day for 12 weeks.
  Interventions: Drug: ORM-12741
- Placebo (Placebo Comparator): Placebo twice a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORM-12741 — ORM-12741 low dose twice a day
  Arms: ORM-12741 low dose
Drug: ORM-12741 — ORM-12741 high dose twice a day
  Arms: ORM-12741 high dose
Drug: Placebo — Placebo twice a day
  Arms: Placebo

SUMMARY:
This study evaluates the effect of ORM-12741 on agitation/aggression symptoms in Alzheimer's disease. Two thirds of the patients will receive ORM-12741 and one third will receive placebo.

DETAILED DESCRIPTION:
ORM-12741 is a potent and selective alpha-2C adrenoceptor (AR)-antagonist. Previous results suggest that the compound may have positive effects on both cognitive and neuropsychiatric symptoms of Alzheimer's Disease. In this study, the effect of ORM-12741 will be evaluated on agitation/aggression symptoms and other neuropsychiatric symptoms. Furthermore, cognition and psychotic and depressive symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) for participation in the study (co-signed by the subject's next of kin or caregiver, or other legally acceptable representative.
* Written IC obtained from a consistently available caregiver informant who is knowledgeable of the subject's condition and its progression and is willing to accompany the subject to all visits and supervise the administration of the study medication.
* Age of 55-90 years (inclusive).
* Male or female subjects with diagnosis of probable Alzheimer's Disease.
* Brain imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) consistent with a diagnosis of Alzheimer's Disease (within 18 months or at screening).
* Mini-mental state examination (MMSE) score between 10-24 (inclusive).
* Clinically significant agitation meeting the International Psychogeriatric Association Provisional Criteria for Agitation in Cognitive Impairment. The agitation symptoms need to have been present for at least 4 weeks before the screening visit.
* Neuropsychiatric Inventory agitation/aggression item score at least 4 at screening visit.

Exclusion Criteria:

* Modified Hachinski Ischemia Score (MHIS) > 4.
* Changes in AChE inhibitor (donepezil, rivastigmine or galantamine) dosing within 2 months prior to screening.
* Changes in memantine dosing within 2 months prior to the screening.
* Changes in antidepressant dosing or addition of another antidepressant medication within 2 months prior to the screening.
* Use of antipsychotics at any dose within 1 month prior to screening.
* Use of benzodiazepines, other than short-acting sleep medications, for night at a maximum of 3 nights/week, within 2 months prior to screening.
* Use of any anticholinergic medication within 2 months prior to screening.
* Current use (within the 30 days prior to screening) of medications with known relevant alpha-2C AR affinity (e.g. mirtazapine, mianserin, clonidine, guanfacine or tizanidine) or with high noradrenaline transporter affinity (reboxetine, venlafaxine or duloxetine).
* Current use of other psychotropic agents, unless the dosing has been stable during the last 2 months prior to the screening.
* Myocardial infarction or other clinically significant ischemic cardiac disease, heart failure, or arrhythmia tendency within the past 2 years.
* Current or history of malignancy within 5 years before screening.
* Suicidal ideation in the 6 months before screening or current suicide risk based on the Colombia-Suicide Severity Rating Scale (C-SSRS) (items 4 and 5 exclusionary) or current risk of suicide based on the investigator's judgement.
* Specific findings in MRI or CT that could in the opinion of the investigator affect cognitive function (such as cortical infarct or silent lacuna in a region known to affect cognition).
* Supine heart rate < 48 bpm or > 100 bpm.
* Systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg after a 5-minute rest.
* Symptomatic orthostatic hypotension.
* QTc-Fridericia (QTcF) repeatedly > 450 ms in males or > 470 ms in females.
* Clinically significantly abnormal thyroid-stimulating hormone (TSH), vitamin B12 or folate serum levels at screening.
* Resides in a skilled nursing facility.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Efficacy on aggression/agitation symptoms measured by Neuropsychiatric Inventory Clinician Rating scale | 12 weeks

SECONDARY OUTCOMES:
Efficacy on aggression/agitation symptoms and overall clinical status measured by Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change | 12 weeks
Efficacy on cognitive symptoms measured by Cognitive Drug Research computerized test battery | 12 weeks
Efficacy on daily living measured by Alzheimer's Disease Co-operative Study - Activities of Daily Living inventory | 12 weeks
Safety measured by assessing adverse events | 12 weeks
Plasma concentrations of ORM ORM-12741, metabolites and possible other Alzheimer's disease medication | 12 weeks
Efficacy on aggression/agitation symptoms measured by Cohen Mansfield Agitation Inventory | 12 weeks
Efficacy on cognitive symptoms measured by Alzheimer's Disease Assessment Scale | 12 weeks
Safety measured by vital signs | 12 weeks
Safety measured by electrocardiogram | 12 weeks
Safety measured by laboratory variables | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, Prof, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland